CLINICAL TRIAL: NCT06391307
Title: The Role of Mesenchymal Stem Cell and Exosome in Treating Pilonidal Sinus Disease in Children: A Prospective Randomized Controlled Trial
Brief Title: The Role of Mesenchymal Stem Cell and Exosome in Treating Pilonidal Sinus Disease in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Azizoğlu (Other)
Collaborators: Necmi Kadıoğlu Hospital (Other)
Responsible Party: Sponsor-Investigator, Mustafa Azizoğlu, Head of Department, Necmi Kadıoğlu Hospital
Organization: Necmi Kadıoğlu Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stem Cell PNS
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pilonidal Sinus; Pilonidal Disease
Keywords: pilonidal sinus disease; Children; wound healing; stem cell; exosome
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crystallized phenol (Active Comparator): In this group, the classic non-operative technique is employed. The pilonidal sinus is debrided under local anesthesia, followed by the injection of crystallized phenol into the wound.
  Interventions: Other: Crystallized phenol
- Crystallized phenol + Exosome (Experimental): In this group, the classic non-operative technique is employed. The pilonidal sinus is debrided under local anesthesia, followed by the injection of crystallized phenol + Exosome into the wound.
  Interventions: Biological: Crystallized phenol + Exosome
- Crystallized phenol + Stem Cell (Experimental): In this group, the classic non-operative technique is employed. The pilonidal sinus is debrided under local anesthesia, followed by the injection of crystallized phenol + Stem cell into the wound.
  Interventions: Biological: Crystallized phenol + Stem Cell
- Crystallized phenol + Exosome + Stem Cell (Experimental): In this group, the classic non-operative technique is employed. The pilonidal sinus is debrided under local anesthesia, followed by the injection of crystallized phenol + Stem cell + Exosome into the wound.
  Interventions: Biological: Crystallized phenol + Exosome + Stem Cell

INTERVENTIONS:
Other: Crystallized phenol — Crystallized phenol + Exosome + Stem Cell
  Other Names: Crystallized phenol will be applied to wound area.
  Arms: Crystallized phenol
Biological: Crystallized phenol + Exosome — Crystallized phenol + Exosome will be applied to wound area.
  Arms: Crystallized phenol + Exosome
Biological: Crystallized phenol + Stem Cell — Crystallized phenol + Stem cell will be applied to wound area.
  Arms: Crystallized phenol + Stem Cell
Biological: Crystallized phenol + Exosome + Stem Cell — Crystallized phenol + Exosome + Stem Cell will be applied to wound area.
  Arms: Crystallized phenol + Exosome + Stem Cell

SUMMARY:
Chronic wounds that fail to heal over extended periods pose a significant financial burden on the healthcare system, underscoring the urgent need to enhance clinical treatments. Among the most promising approaches are stem cell-based therapies. Substantial evidence suggests that mesenchymal stem cells (MSCs) can facilitate the healing of chronic wounds in both animal models and preclinical studies, primarily through their paracrine actions. The bioactive factors and cytokines secreted by MSCs can be harvested in the form of conditioned medium. This medium has been processed into a lyophilized powder for clinical use. Patients with chronic wounds will recruited and divided into two groups: the control group will receive the commonly used fibroblast growth factor, while the experimental group was treated with the lyophilized powder. The study aims to assess the efficacy and safety of this Stem cell and exosome in treating chronic wounds (especially pilonidal sinus).

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is an infectious or inflammatory condition beneath the skin at the peak of the gluteal cleft in the sacrococcygeal area. It is a chronic condition characterized by discharge, infection, and pain. Although it can occur during adolescence, it is most commonly seen in adult males, leading to a focus on adult treatments in research. Surgical treatment was first implemented by Anderson in 1847. Since then, various surgical and medical treatment options have been explored, yet there is no widely accepted standardized treatment. The ideal treatment should be simple, require a short hospital stay, have low recurrence rates, provide good cosmetic results, be cost-effective, cause minimal pain, and allow a quick return to social life, making the surgical approach contentious.

Maurice and Greenwood first reported the application of liquid phenol in 1964, initially under general anesthesia, later shifting to local anesthesia. Due to high recurrence rates with liquid phenol, Dogru and colleagues introduced the crystallized phenol (CP) procedure, a minimally invasive method now commonly used in adults.

Recent years have shown that stem cells and exosomes promote tissue healing and reduce inflammation. Known for their ability to differentiate into various cell types, stem cells, and exosomes play critical roles in intercellular communication, containing a variety of molecules. Their use in surgical fields has become popular as they speed up the post-operative healing process and reduce the risk of complications. Research in the literature supports that stem cells and exosomes accelerate wound healing (e.g., Nourian Dehkordi A, et al. 2019).

This study is based on two main premises: firstly, to identify the potential healing effects of stem cell and exosome applications in treating pilonidal sinus disease; and secondly, to comparatively assess the impact of these applications on surgical outcomes, specifically regarding surgery duration, complications, and the healing process. Comparing these two groups will help determine the value of stem cell and exosome applications in managing pilonidal sinus disease.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years children.
* Patients with chronic non-healing wound and pilonidal sinus diseases.

Exclusion Criteria:

* Patients with epilepsia
* Patients with diabetes
* Patients with hypertension
* Patients with chronic other diseases.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | 3 weeks
  In the control group, the healing process generally takes about 2-3 weeks. In the experimental group, a shorter duration is expected. In this study, the wound healing times of both groups will be evaluated and compared.
Cosmetic results | 2 month
  In this study, the worst healing wounds will receive a score of 1, and the best-healed wounds, which are closest to normal skin, will receive a score of 10. In short, a low score indicates poor wound healing and poor cosmetic, while a high score indicates that the wound has achieved a good cosmetic appearance.
Skin burn rate | 2 weeks
  In patients treated with crystallized phenol, skin burns can occur during application. To prevent this, Furacin ointment is applied around the wound. However, we still encounter skin burns. In this study, it is expected that the experimental groups will have a lower burn rate compared to the control group. The burn rate will be evaluated in this study.
Average time to full daily activities | 1 week
  It refers to the time when patients return to their routine lives after the procedure.
VAS score | 7 weeks
  Patient visual analog scale (VAS) scores will be assessed both prior to the procedure and again 10 days, 20 days following the procedure and after recovery.
Success rate | 7 weeks
  The succes rate will be calculated after interventions
Recurrence rate | 7 weeks
  The recurrence rate will be calculated after interventions

SECONDARY OUTCOMES:
Bleeding rate | 1 week
  Bleeding during interventions will be calculated
Infection rate | 7 week
  Infection will be defined during interventions and 10 days after intervention
Total complication rate | 7 weeks
  Total complicaitons during interventions will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoğlu, MD, Principal Investigator — Esenyurt State Hospital
Locations (1):
- Mustafa Azizoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No